CLINICAL TRIAL: NCT03076164
Title: A Phase 1/2 Trial of Trametinib and Erlotinib in Patients With EGFR-Mutant Lung Adenocarcinomas and Acquired Resistance to Erlotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-098
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2020-06

CONDITIONS: Lung Adenocarcinoma; Lung Cancer; Lung Cancer Metastatic; Lung Cancer Stage IV; Recurrent Lung Adenocarcinoma; Recurrent Lung Cancer
Keywords: erlotinib; trametinib; 15-098
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — trametinib; Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: Trametinib 1.5mg + Erlotinib 75mg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trametinib 1.5mg + Erlotinib 75mg (Experimental): Phase 1: Accrue 6 patients on Trametinib 1.5mg + Erlotinib 75mg by mouth once daily Phase 2: Accrue 24 patients (including 6 patients treated during Phase 1) on Trametinib 1.5mg + Erlotinib 75mg by mouth once daily or Trametinib 1.0mg + Erlotinib 100mg by mouth once daily.
  Interventions: Drug: Trametinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Trametinib — Trametinib 1.5mg once daily by mouth
Drug: Erlotinib — Erlotinib 75mg once daily by mouth

SUMMARY:
The purpose of this study is to determine the safety, tolerability and overall response rate of trametinib when given in combination with erlotinib in patients with Stage IV or recurrent lung adenocarcinoma that cannot be treated with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of advanced stage IV or recurrent lung adenocarcinoma reviewed at MSKCC
* Somatic activating mutation in EGFR Radiographic progression during treatment with erlotinib.
* Any number of prior chemotherapy regimens is permitted.
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* KPS >/= 70%
* Age >18 years old
* Must have undergone biopsy after development of acquired resistance to erlotinib with available archived tissue (equivalent of > 10 unstained slides)
* Left ventricular Ejection Fraction >/= the lower limit of normal by ECHO or MUGA
* Adequate organ function:
* AST, ALT </= 2.5 x ULN
* Total bilirubin </= 1.5 x ULN
* Albumin>/=2.6g/dL - Creatinine < 1.5 x ULN OR calculated creatinine clearance >/=50mL/min
* Absolute neutrophil count (ANC) >/= 1,200 cells/mm3
* Hemoglobin>/=9.0 g/dL
* Platelets >/=100,000/mm3

Exclusion Criteria:

* Patients with symptomatic brain metastasis requiring escalating doses of steroids
* Patients with grade 2 or greater diarrhea prior to study initiation despite maximal medical management due to medications or a medical condition such as Crohn's disease or malabsorption
* Pregnant or lactating women
* Any type of systemic therapy (chemotherapy or experimental drugs) within 2 weeks of starting treatment on protocol except for a EGFR TKI
* Patients who have received prior treatment with a MEK inhibitor
* Any major surgery or extensive radiotherapy within 21 days of starting treatment on protocol.
* A history of clinically significant interstitial lung disease or pneumonitis
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study administration, New York Heart Association Class III or IV congestive heart failure, or symptomatic uncontrolled Arrythmias, prolonged corrected QT interval >480msec, treatment refractory hypertension, presence of a cardiac defibrillator
* History of central serous retinopathy or retinal vein occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This treatment regimen was already assessed in a previous study. The phase 1 portion was a safety lead-in of a slight modification of the previously established combination dosing. As a consequence, we only did a safety lead in of one dose level that was determined to be the phase 2 dose and we rolled all the phase 1 patients into the phase 2 cohort.
Groups:
- Trametinib 1.5mg + Erlotinib 75mg: Phase 1: Accrue 6 patients on Trametinib 1.5mg + Erlotinib 75mg by mouth once daily Phase 2: Accrue 24 patients (including 6 patients treated during Phase 1) daily doses of 75mg erlotinib and 1.5mg trametinib
  This treatment regimen was already assessed in a previous study. The phase 1 portion was a safety lead-in of a slight modification of the previously established combination dosing. As a consequence, we only did a safety lead in of one dose level that was determined to be the phase 2 dose and we rolled all the phase 1 patients into the phase 2 cohort. There would be no reason or utility to assess the phase 1 cohort separately since they received the same dose as the phase 2 cohort.
Period: Overall Study
Arm/Group | Trametinib 1.5mg + Erlotinib 75mg
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Trametinib 1.5mg + Erlotinib 75mg: Phase 1: Accrue 6 patients on Trametinib 1.5mg + Erlotinib 75mg by mouth once daily Phase 2: Accrue 24 patients (including 6 patients treated during Phase 1) daily doses of 75mg erlotinib and 1.5mg trametinib This treatment regimen was already assessed in a previous study. The phase 1 portion was a safety lead-in of a slight modification of the previously established combination dosing. As a consequence, we only did a safety lead in of one dose level that was determined to be the phase 2 dose and we rolled all the phase 1 patients into the phase 2 cohort.
Arm/Group | Trametinib 1.5mg + Erlotinib 75mg
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Participants Response Rate
Description: Response and progression of disease will be evaluated in this study using interval imaging every 8 weeks with CT scan of the chest and imaging of any other target lesion with response evaluated by RECIST 1.1.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Trametinib 1.5mg + Erlotinib 75mg
Number analyzed (Participants) | 24
participants
  Stable Disease | 11
  Progression of disease | 4
  Not Entered | 8
  Partial Response | 1

2. Primary Outcome: Number of Participants Evaluated for Toxicities
Description: Safety and tolerability will be evaluated by systematic and regular toxicity evaluations. Toxicity will be graded according to NCI CTCAE version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Trametinib 1.5mg + Erlotinib 75mg
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Trametinib 1.5mg + Erlotinib 75mg
All-Cause Mortality (participants affected / at risk) | 20/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib 1.5mg + Erlotinib 75mg (N=24)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Malaise (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib 1.5mg + Erlotinib 75mg (N=24)
Diarrhea (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 15
Rash acneiform (Skin and subcutaneous tissue disorders) | 13
Nausea (Gastrointestinal disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Aspartate aminotransferase increased (Investigations) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Alanine aminotransferase increased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 4
Edema limbs (General disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Fever (General disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Skin infection (Infections and infestations) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Gen disorders & admin site conditions Other, spec (General disorders) | 2
Malaise (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Rectal hemmorhage (Gastrointestinal disorders) | 2
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03076164/Prot_SAP_000.pdf